CLINICAL TRIAL: NCT07071207
Title: Effect of Text Message Reminders on Michigan Incontinence Symptom Index Score After Prostate Surgery
Brief Title: Effect of Text Message Reminders on M-ISI Score After Prostate Surgery
Acronym: TextMsgM-ISI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Scott Quarrier, Assistant professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00009182
Record Dates: First submitted 2025-03-07; First posted 2025-07-17 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Incontinence, Urinary Stress; Prostate Cancer; Benign Prostate Hyperplasia
MeSH Terms: conditions — Urinary Incontinence, Stress; Prostatic Neoplasms; Prostatic Hyperplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control group - LEP surgery patients (No Intervention): Patients undergoing LEP surgery and standard of care discharge instructions to perform pelvic floor exercises
- Intervention group - LEP surgery patients (Experimental): Patient undergoing LEP surgery with text message intervention to perform pelvic floor exercises as described in the schedule of events
  Interventions: Behavioral: Text message reminders
- Control group - RALP surgery patients (No Intervention): Patients undergoing RALP surgery and standard of care discharge instructions to perform pelvic floor exercises
- Intervention group - RALP surgery patients (Experimental): Patient undergoing RALP surgery with text message intervention to perform pelvic floor exercises as described in the schedule of events
  Interventions: Behavioral: Text message reminders

INTERVENTIONS:
Behavioral: Text message reminders — daily 8am text messages reminding patients to perform Kegel exercises as per their standard-of-care post-operative discharge instructions.
  Arms: Intervention group - LEP surgery patients; Intervention group - RALP surgery patients

SUMMARY:
The purpose of this study is to compare post-prostatectomy incontinence via Michigan Incontinence Score Index in patients receiving daily text message reminders for pelvic floor exercises when compared to those not receiving text reminders.

DETAILED DESCRIPTION:
This trial will be comprised of prostate cancer patients who have undergone a radical prostatectomy and benign prostate hyperplasia patients who have undergone a laser enucleation of the prostate. These two cohorts will each be split into an intervention and a control group. The purpose of this study is to evaluate post-prostatectomy incontinence via patient reported outcomes utilizing Michigan Incontinence Score Index in patients receiving daily text message reminders for pelvic floor exercises + standard of care (intervention group) compared to those receiving standard of care only (control group).

ELIGIBILITY:
Inclusion Criteria:

1. Planning to undergo a radical prostatectomy (RALP) or laser enucleation of the prostate (LEP) procedure
2. Patient of URMC Urology
3. Adult male 18 years of age and older
4. Able to read, write, and speak in English (NOTE: due to limitations with questionnaire validation, only English-speaking subjects are permitted)
5. Has access to a mobile device capable of receiving automated text messages.
6. Willing to receive text messages and to complete questionnaires via SMS text.
7. Willingness to participate and able to provide informed consent.

Exclusion Criteria:

1. Less than 18 years of age
2. Unable to send and receive SMS texts
3. Unable to read, write, and speak English
4. Catheter dependency
5. Has or plans to have Artificial Urinary Sphincter or Urethral Sling during the study period
6. In the opinion of the investigator, the subject has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2025-09-15 (Actual); Primary Completion 2028-05-01 (Estimated); Study Completion 2028-05-01 (Estimated)

PRIMARY OUTCOMES:
Time to Recovery to Continence | From baseline until the participant reaches two successive M-ISI Pad Use Subdomain Scores of ≤ 2, assessed up to 12 months
  The time it takes for participants to recover continence, as defined by two successive M-ISI Pad Use Subdomain Scores of ≤ 2. The Pad Use Subdomain Score is determined by the sum of items Q7-8 from the M-ISI questionnaire, assessed as a time-to-event outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- 158 Sawgrass clinic; Suite 3100, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No